CLINICAL TRIAL: NCT06176001
Title: Group-based Psychoeducation for Relatives of Patients With Bipolar Disorder - a Large Scale Real-world Randomized Controlled Parallel Group Trial
Brief Title: Group-based Psychoeducation for Relatives of Patients With Bipolar Disorder, a Randomized Controlled Trial
Acronym: R-Bipolar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Principal Investigator, Lars Vedel Kessing, professor, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P-2021-809
Record Dates: First submitted 2023-11-29; First posted 2023-12-19 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-06

CONDITIONS: Bipolar Disorder
Keywords: Relatives; Caregivers; Family; Psychoeducation; Randomized controlled trial
MeSH Terms: conditions — Bipolar Disorder | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psychoeducation (Active Comparator): Participants randomized to this arm are offered group-based psychoeducation shortly thereafter.
  Interventions: Other: psychoeducation in groups
- Waiting list (Placebo Comparator): Participants randomized to this arm are placed on a waiting list for approximately 4 months and then offered group-based psychoeducation thereafter.
  Interventions: Other: psychoeducation in groups

INTERVENTIONS:
Other: psychoeducation in groups — Group-based psychoeducation for relatives. Group size: 20-40 relatives. Duration of intervention: six sessions, each two hours long with a 15 minutes break, over a period of 6-10 weeks. The sessions are held by experienced clinicians from the Copenhagen Affective Disorder Clinic, one chief physician and one nurse. Each session focuses on a specific topic, which the clinicians present and discuss using a presentation viewer. The sessions are interactive, and the participants are encouraged to ask questions during the presentations. During each session the participants will have some discussions in smaller groups to reflect on a topics and issues raised during the session.

SUMMARY:
Relatives of patients with bipolar disorder (BD) often experience emotional burden with stress, and depressive symptoms that again increases the likelihood of destabilization and relapses in the patient. The effects of group-based psychoeducation have not been investigated in large-scale real-world settings. The investigators are currently conducting a large-scale real-world randomized controlled parallel group trial (RCT) to test whether group-based psychoeducation for relatives to patients with BD improves mood instability and other critical outcomes in relatives and the corresponding patients with BD.

The trial is designed as a two-arm, parallel group randomized trial with a balanced randomization 1:1 to either group-based psychoeducation or a waiting list for approximately 4 months and subsequent group-based psychoeducation. the investigators plan to include 200 relatives. The group sizes for psychoeducation is between 20-40 relatives.The primary outcome measure is mood instability calculated based on daily smartphone-based mood self-assessment. Other relevant outcomes are measured, including patients' reported outcomes, assessing self-assessed burden, self-efficacy, and knowledge about BD.

ELIGIBILITY:
Inclusion Criteria:

* Relatives of patients with Bipolar Disorder who are affiliated with the Copenhagen Affective Disorder Clinic.

Exclusion Criteria:

* Insufficient Danish language.
* Age below 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in mood instability in the relatives | daily in 4-8 months.
  Mood instability is calculated from daily self-reported mood registration in the app Monsenso. Participating relatives score their daily mood on a 9-point scale from 0-8 where 8 is 'in a brilliant mood' and 0 is 'really sad'
  The participant rate daily in the Monsenso app during the time the participate in the study (4-8 months depending on which group they are randomly allocated to).
  For each participant, a mood instability measure will be estimated for each day and aggregated by applying the root mean square successive difference (rMSSD) method.
Change in mood instability in the corresponding patients | daily in 4-8 months.
  Mood instability is calculated from daily self-reported mood registration via the app Monsenso. The patients score their daily mood on a scale from -3 to +3, where -3 is the worst and +3 is the best mood. Patients' data from the Monsenso app is collected from a parallel RCT, in the time frame in which the relatives are in the study.

SECONDARY OUTCOMES:
Self-reported daily registrations in the Monsenso app on the following topics: daily activity level, sleep, mixed moods, anxiety, irritability, cognition, stress, alchohol consumption, patient support and level of burden from being a caregiver, | daily 4-8 months.
  Each topic is covered by a single, simple question in the Monsenso app:
  * Daily activity level: 'how active have you been?' (7-point scale from very little to very much)
  * Sleep: How many hours did you sleep (scale from 0 to 12+hours)
  * mixed moods: have you experienced mixed good and bad mood? (yes/no)
  * Anxiety: Have you felt anxiety? (5-point scale from 'not at all' to 'to a high degree')
  * Irritability:Have you felt irritable? (5-point scale, same as above)
  * Cognition: Have you experienced cognitive difficulties? (5-point scale, same as above)
  * Stress: Have you been stressed? (5-point scale, same as above)
  * Alcohol: how many drinks have you had? (scale from 0 til 10+ drinks)
  * Patient support: Have you helped or supported the patient? (5-point scale, same as above)
  * Caregiver burden: To which degree have you experienced the patient's mental health problems as a burden to you? (5-point scale, same as above)
Self-rated caregiver burden | at inclusion, at follow-up around 4 months, and if in control group at around 7-8 months
  Burden Assessment Scale
  19 questions covering subjects as economic and practical burden, stigma, worries, conflicts etc, participants answer on a scale from [1: not at all] to [4: to a high degree] or [not relevant]
  Reinhard SC, Gubman GD, Horwitz AV, Minsky S. Burden assessment scale for families of the seriously mentally ill. Eval Program Plann. 1. juli 1994;17(3):261-9.
Self-rated expressed emotions | at inclusion, at follow-up around 4 months, and if in control group at around 7-8 months
  Perceived Criticism Measure
  The questionnaire consists of four questions covering criticism in a relationship, answered on a scale from 0 to 10, where 10 is the highest and most negative.
  Hooley JM, Parker HA. Measuring expressed emotion: An evaluation of the shortcuts. J Fam Psychol. september 2006;20(3):386-96.
Self-rated quality of life | at inclusion, at follow-up around 4 months, and if in control group at around 7-8 months
  Carer Quality of Life
  7 multiple-answer questions and one Visual Analog Scale to evaluate quality of life in the light of being an informal caregiver.
  Brouwer WBF, van Exel NJA, van Gorp B, Redekop WK. The CarerQol instrument: A new instrument to measure care-related quality of life of informal caregivers for use in economic evaluations. Qual Life Res. 1. august 2006;15(6):1005-21.
  Hoefman RJ, van Exel NJA, Looren de Jong S, Redekop WK, Brouwer WBF. A new test of the construct validity of the CarerQol instrument: measuring the impact of informal care giving. Qual Life Res. 2011;20(6):875-87.
Self-rated carer self-efficacy | at inclusion, at follow-up around 4 months, and if in control group at around 7-8 months
  Carer-Self-Efficacy
  12 questions about self-efficacy as a caregiver for a person with Bipolar disorder. The questionnaire was originally developed for persons with bipolar disorder (Smith) and later Hubbard et al made a version for caregivers.
  Smith LM, Erceg-Hurn DM, McEvoy PM, Lim L. Self-efficacy in bipolar disorder: Development and validation of a self-report scale. J Affect Disord. 1. februar 2020;262:108-17.
  Hubbard AA, McEvoy PM, Smith L, Kane RT. Brief group psychoeducation for caregivers of individuals with bipolar disorder: A randomized controlled trial. J Affect Disord. august 2016;200:31-6.
Knowledge about bipolar | at inclusion, at follow-up around 4 months, and if in control group at around 7-8 months
  25 questions testing the factual knowledge about bipolar disorder.
  "The Bipolar disorders knowledge scale", Trevor A. Stump and Marty L. Eng. Journal of Affective disorders, 2018-10-01, Volume 238, Pages 645-650.
Self-rated health related quality of life | at inclusion, at follow-up around 4 months, and if in control group at around 7-8 months
  Short Form-12 (54,55) 12 questions on health-related quality of life.
  Christensen LN, Ehlers L, Larsen FB, Jensen MB. Validation of the 12 Item Short form Health Survey in a Sample from Region Central Jutland. Soc Indic Res. 1. november 2013;114(2):513-21.
  Amir M, Lewin-Epstein N, Becker G, Buskila D. Psychometric properties of the SF-12 (Hebrew version) in a primary care population in Israel. Med Care. oktober 2002;40(10):918-28.
Self-rated mental health | at inclusion, at follow-up around 4 months, and if in control group at around 7-8 months
  The Brief Symptom Inventory (BSI: Derogatis, 1992), a 53-item self-report inventory of psychopathology and psychological distress, the BSI psychometric profile produces the same nine primary symptom dimensions produced by the SCL-90-R.
  Derogatis LR, Melisaratos N. The Brief Symptom Inventory: an introductory report. Psychol Med. august 1983;13(3):595-605.
Self-rated stress | at inclusion, at follow-up around 4 months, and if in control group at around 7-8 months
  Perceived Stress Scale
  10 questions covering stress symptoms in the last month.
  Cohen S. Perceived stress in a probability sample of the United States. I: The social psychology of health. Thousand Oaks, CA, US: Sage Publications, Inc; 1988. s. 31-67. (The Claremont Symposium on Applied Social Psychology).
Self-rated bipolar symptoms | at inclusion, at follow-up around 4 months, and if in control group at around 7-8 months
  Mood Disorder Questionnaire
  Hirschfeld RMA, Williams JBW, Spitzer RL, Calabrese JR, Flynn L, Keck PE, m.fl. Development and Validation of a Screening Instrument for Bipolar Spectrum Disorder: The Mood Disorder Questionnaire. Am J Psychiatry. november 2000;157(11):1873-5.
Self-rated depressive symptoms | at inclusion, at follow-up around 4 months, and if in control group at around 7-8 months
  Major Depression Inventory
  Bech P, Timmerby N, Martiny K, Lunde M, Soendergaard S. Psychometric evaluation of the Major Depression Inventory (MDI) as depression severity scale using the LEAD (Longitudinal Expert Assessment of All Data) as index of validity. BMC Psychiatry. 5. august 2015;15:190.
  Bech P, Wermuth L. Applicability and validity of the Major Depression Inventory in patients with Parkinson's disease. Nord J Psychiatry. (52):305-10.
Self-rated Childhood trauma | Only at inclusion
  Childhood Trauma Questionnaire (CTQ)
  Bernstein DP, Fink L, Handelsman L, Foote J, Lovejoy M, Wenzel K, m.fl. Initial reliability and validity of a new retrospective measure of child abuse and neglect. Am J Psychiatry. august 1994;151(8):1132-6.
Clinically observer rated Depressive symptoms | At inclusion, at 3-4 months and for the control-group also at 7-8 months.
  Depressive symptoms assessed by the Hamilton Depression Rating Scale-6 items (min. value = 0; max. value = 22, with higher values reflecting more depressive symptoms)
  Hamilton M. A rating scale for depression. J Neurol Neurosurg Psychiatry. februar 1960;23(1):56-62.
Clinically observer rated Manic symptoms | at inclusion, at follow-up around 4 months, and if in control group at around 7-8 months
  Manic symptoms assessed by the Young Mania Rating Scale (min. value = 0; max. value = 60, with higher values reflecting more manic symptoms)
  Young RC, Biggs JT, Ziegler VE, Meyer DA. A rating scale for mania: reliability, validity and sensitivity. Br J Psychiatry J Ment Sci. november 1978;133:429-35.
Clinically observer rated General functioning | at inclusion, at follow-up around 4 months, and if in control group at around 7-8 months
  General functioning assessed by the Functional Assessment Short Test, a 24-item interviewer-administered interview concerning autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships and leisure time (min. value = 0; max. value = 72, with higher values reflecting poorer function)
  Rosa AR, Sánchez-Moreno J, Martínez-Aran A, Salamero M, Torrent C, Reinares M, m.fl. Validity and reliability of the Functioning Assessment Short Test (FAST) in bipolar disorder. Clin Pract Epidemiol Ment Health CP EMH. 7. juni 2007;3:5.

OTHER OUTCOMES:
Change in automatically smarthone-generated data | 4-8 months
  Automatically smartphone-generated data on physical - and social activity is generated in the Monsenso app using the phone's sensor-data.
  physical activity: location and physical activity (step count and movement) social activity: battery level, light level and screen mode.
  These automatically generated data has been shown to be informative in prior study:
  Faurholt-Jepsen M, Frost M, Vinberg M, Christensen EM, Bardram JE, Kessing LV. Smartphone data as objective measures of bipolar disorder symptoms. Psychiatry Res. 30. juni 2014;217(1-2):124-7.

CONTACTS AND LOCATIONS:
Overall Officials: Lars V Kessing, professor, Principal Investigator — Copenhagen Psychiatric Center
Locations (1):
- Copenhagen Affective Disorder Clinic, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stokholm JR, Waldemar AK, Kessing LV. Becoming diplomats with boundaries - a thematic analysis of relatives' experiences with group-based psychoeducation about bipolar disorder. BMC Psychiatry. 2025 Sep 1;25(1):843. doi: 10.1186/s12888-025-07219-y. PMID 40890647
- [Derived] Stokholm JR, Vinberg M, Faurholt-Jepsen M, Kessing LV. Study protocol: group-based psychoeducation for relatives of patients with bipolar disorder-a large scale real-world randomized controlled parallel group trial, the R-bipolar RCT. Trials. 2024 May 23;25(1):342. doi: 10.1186/s13063-024-08172-z. PMID 38783322